CLINICAL TRIAL: NCT05109429
Title: Developing a Clinical Outcome Assessment for Opioid Craving
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00302133; R21DA054952 (NIH)
Record Dates: First submitted 2021-10-15; First posted 2021-11-05 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Opioid Craving; Opioid Use Disorder; Measure Development
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will experience all three cue-induced craving tasks (no, low, and high) in a random order (6 possible orders)
Masking Description: It is not possible to blind the participant nor some of the research staff to the study condition. The research staff who will interview the participant will be blinded to what cue condition participant had completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No Craving (Experimental): Each participant will attend three sessions where the participant will experience three distinct cue-induced craving tasks in a randomized fashion.
  Interventions: Behavioral: Neutral Cue-induced Craving; Behavioral: Visual Opioid Cue-induced Craving; Behavioral: Visual and Tactile Opioid Cue-induced Craving

INTERVENTIONS:
Behavioral: Neutral Cue-induced Craving — For the neutral cue condition, the participant will be seated in front of a 16-inch monitor and instructed to sit upright to view 20 pictures of water bottles via E-Prime software (Psychology Software Tools Inc., PA), presented for five seconds each in randomized order. The images will include pictures of a water bottle alone, water being poured from a bottle to a glass, and an individual drinking from a bottle of water. Next, participants will watch as research staff open a bottle of water, pour it into a glass, and place it on a table in front of the participant. Participants will also be asked to look at a water bottle, hold it, sniff it, and take a drink of water.
Behavioral: Visual Opioid Cue-induced Craving — For the visual opioid cue-induced craving condition, the participant will again be seated in front of a 16-inch monitor and instructed to sit upright to view 20 pictures of opioid-related imagery, presented for five seconds each in a randomized order. The opioid-related imagery will be customized for heroin or prescription opioids based upon the participant's primary opioid of choice. The images will include pills and white powder, stages of drug taking preparation (e.g., holding spoon over flame, pills being crushed).
Behavioral: Visual and Tactile Opioid Cue-induced Craving — For the visual and tactile opioid cue condition, procedures will differ depending on the participants' most preferred route of administration. . Intranasal users will be instructed to watch as research staff opens a wallet, removes a $1 bill, removes a packet of powder mimicking heroin/crushed pills, open the packet, and roll the dollar bill. The participant will then be given the packet and the dollar bill to hold for approximately 30 seconds. Intravenous users will be instructed to watch the research nurse open the packet of fake heroin, pour its contents into a spoon, added a few drops of water to the spoon, hold an open flame from a lighter under the spoon, add cotton to the spoon, and draw the fluid into a syringe.

SUMMARY:
The purpose of this study is to collect information about opioid craving so that the investigators can develop an opioid craving assessment to improve treatments for individuals with opioid use disorder. To collect this information, the investigators are recruiting individuals in treatment for opioid use disorder who will complete cue-induced opioid craving tasks where these individuals will: (1) look at pictures of neutral objects and touch neutral objects (e.g., water bottles or flashlights), (2) look at opioid-related images, and (3) look and touch opioid-related objects. Participants will then complete a one-on-one interview about the thoughts, feelings and physical sensations the participants experienced during the cue-induced craving session. Participants will also complete questionnaires and existing opioid craving assessments. Finally, participants will provide formal feedback about existing opioid craving assessments with cognitive interviews.

DETAILED DESCRIPTION:
There is no universally accepted and validated assessment for opioid craving. Craving is a symptom among individuals with opioid use disorder which can contribute to instances of relapse. More research is needed to develop a valid opioid craving assessment which captures all relevant opioid craving dimensions. Developing a valid, FDA-qualified assessment would support the creation of novel interventions to treat opioid craving and facilitate FDA labeling of a treatment for mitigating opioid craving. To establish content validity, the FDA requires (1) qualitative feedback from stakeholder populations about what should be included in an assessment of opioid craving, and (2) standardized interviews which evaluate participant's acceptability and comprehension of existing assessments of opioid craving. The investigators propose collecting qualitative data in a rigorous laboratory model of cue-induced opioid craving to establish content validity for a craving assessment. Participants (n = 81) will be individuals who are in treatment for opioid use disorder. Participants will attend three outpatient laboratory sessions where the participants will be separately exposed to (1) visual and tactile neutral cues, (2) visual opioid cues, and (3) visual and tactile opioid cues; corresponding to "no", "low", and "high" levels of cue-induced craving. Following cue exposure, participants will be asked to describe in participants' own words the thoughts, moods, and symptoms the participants experience during and after the cue-induced craving task. Next, participants will be asked to complete a brief symptom checklist and rate participants' level of craving for opioids on 9 existing craving questions. Participants will also be asked to provide feedback on existing craving assessments in a standardized interview. Ultimately, these data will identify craving domains experienced across relevant stakeholder populations during both low and high craving bouts.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Opioid-positive urine sample at admission visit (excluding individuals receiving Naltrexone).
* Current opioid use disorder per Diagnostic Statistical Manual (DSM)-5
* Currently in treatment for opioid use disorder

Exclusion Criteria:

* Being pregnant or breastfeeding, or may become pregnant during the trial
* History of psychosis or mania or other serious psychiatric disorders assessed by the Mini International Neuropsychiatric Interview
* Past 30-day suicidal behavior assessed by the Columbia Suicide Severity Rating Scale
* Have circumstances that would interfere with study participation (e.g., impending jail).
* Positive for illicit substances except opioids and cannabis
* Current substance use disorder other than opioid or nicotine
* Current intoxication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Craving Domains | Sessions 1, 2, and 3 after the cue-induced craving task (approximately 1 hour into session)
  Immediately following each cue condition, participants will be asked the following open-ended questions: (1) Describe your mood, (2) Describe how you feel, and (3) What symptoms are you experiencing? Responses will be recorded using a digital audio recorder.
  Qualitative data collected on the symptoms, moods and feelings following cue-induced craving tasks will be transcribed and independently coded for common craving domains based on our published preliminary study by two raters. Raters will also document other potential domains that do not fit into any of the a priori categories. Ad Hoc domains require that both raters agree that a new category should be created. Independently coded responses will be compared and incongruencies will be reviewed by a third rater who will make the final designation. The types and frequencies of craving domains will be summarized with descriptive statistics.
Change in Acceptability of Craving Assessments | Sessions 1, 2, and 3 after cue-induced craving task (approximately 1 hour into session)
  Responses to the question "What was this question designed to measure?" will be coded by two independent raters as either "Demonstrates understanding" or "Does not demonstrate understanding". Next, responses to the question "What would you change, if anything, about this measure?", will be transcribed and independently coded by two raters as either "no changes needed" or "changes needed". Responses will be compared and incongruencies will be reviewed by a third rater who will make the final designation. If final responses to either question is determined to be either "does not demonstrate understanding" and/or "changes needed", the question will be labeled as unacceptable. For each craving assessment item, the proportion of participants who describe the item as unacceptable will be computed. The proportions of responses designated as "does not demonstrate understanding" and "changes needed" will also be computed.
Change in Deficits in Craving Assessments | Sessions 1, 2, and 3 after cue-induced craving task (approximately 1 hour into session)
  Responses to the question "What was not captured by these questions that you would include in a measure for assessing opioid craving?" will be coded for themes by two independent raters. Independently coded responses will be compared and incongruencies will be reviewed by a third rater who will make the final designation. The types and frequencies of recommendations will be summarized with descriptive statistics.

SECONDARY OUTCOMES:
Change in Predictive utility of craving assessment items | Sessions 1, 2, and 3 during and immediately after the cue-induced craving assessment (approximately 1 hour into session)
  Average measures of heart rate and galvanic skin response 10 minutes prior to cue-exposure will be subtracted from average measures of heart rate and galvanic skin response for the 10 minutes beginning with cue-exposure to calculate a change from baseline measure of both physiological measures. Greater changes will be indicative of a greater conditioned response. (1) Logistic mixed effects models will evaluate the association between change from baseline physiological measures and whether an individual described a given craving domain across craving condition (domain present, domain absent) and stakeholder group . (2) Linear mixed effects models will evaluate the association between change from baseline heart rate and galvanic skin response and scores on existing craving question single item scores (range: 0-100 and 0-9) across craving condition and stakeholder group. Greater scores on single item craving questions are associated with greater craving.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia L Bergeria, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No